CLINICAL TRIAL: NCT02779712
Title: Remote Ischaemic Conditioning After Stroke Trial (ReCAST-2): A Pilot Randomised Controlled Phase II Trial Evaluating Remote Ischaemic Conditioning (RIC) After Hyperacute Stroke 2
Brief Title: Remote Ischaemic Conditioning After Stroke Trial (ReCAST-2)
Acronym: ReCAST-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16007
Record Dates: First submitted 2016-01-22; First posted 2016-05-20 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2017-07

CONDITIONS: Stroke
Keywords: Remote ischaemic conditioning
MeSH Terms: conditions — Stroke | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remote Ischaemic Conditioning (Active Comparator): Remote ischaemic conditioning (RIC group): 4 cycles of intermittent limb ischaemia - alternating 5 minutes inflation (20mmHg above systolic BP) followed by 5 minutes deflation of a standard upper arm blood pressure cuff
  Interventions: Procedure: Remote ischaemic conditioning
- Control (Sham Comparator): Control: 4 cycles of alternating 5 minutes inflation (up to 30 mmHg) followed by 5 minutes deflation of a standard upper arm blood pressure cuff
  Interventions: Procedure: Sham

INTERVENTIONS:
Procedure: Remote ischaemic conditioning — 1 dose (=4 cycles) of intermittent upper limb ischaemia (1 cycle = 5minutes inflation to 20mmHg above systolic BP, 5 minutes deflation). Dose escalation: (i) Recruits 1-20 receive this cycle once (ii) Recruits 21-40 receive a second dose of 4-cycles one hour after the first. (iii) Recruits 41-60 receive further dosing, twice daily until day 4.
  Arms: Remote Ischaemic Conditioning
Procedure: Sham — 4 cycles of intermittent sham procedure (1 cycle = 5 minutes inflation to 30 mmHg, 5 minutes deflation), matching the dose escalation described in the intervention
  Arms: Control

SUMMARY:
Stroke has an enormous impact on both individual and society. Novel treatments are required to relieve this burden and remote ischaemic conditioning (RIC) is one such approach. RIC refers to applying non-lethal ischaemia to an area distant from an organ you are trying to protect (e.g. the brain). Pre-clinical animal stroke studies have shown RIC to be neuroprotective and help restore functional outcome when compared to control. These outcomes are achieved simply by transiently occluding the blood supply to a limb (e.g. the arm) very soon after the stroke occurs. The mechanisms of protection are unclear but may be due enhancing the body's ability to protect itself from further injury by favorably altering cerebral blood flow or reducing the detrimental effects of oxygen free radicals. Ischaemic conditioning (IC) is an intervention already applied during cardiac surgery to protect the heart from damage and it may be effective after an acute myocardial infarction. The investigators therefore plan to conduct a pilot randomised controlled trial assessing the feasibility of applying RIC (4 cycles of blood pressure cuff inflation for 5 minutes) in patients within 6 hours of ischaemic stroke. The primary outcome is feasibility of RIC. Secondary outcomes include tolerability, safety and clinical efficacy. The results will inform the design of future trials of a potential intervention is that is pragmatic, non-invasive and simple to administer.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected clinical stroke with 6 hours of onset of neurological symptoms;
2. Age >18;
3. Written or witnessed oral consent, or relative/consultee advice.

Exclusion Criteria:

1. Pre-morbid dependency mRS>3;
2. Dementia;
3. Coma (GCS< 8);
4. Malignancy or significant co-morbidity thought to limit life expectancy to <6 months;
5. Blood sugar < 3.5 mmol/L;
6. Taking part in another clinical trial of an investigational medicinal product (CTIMP);
7. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-07-23 (Actual); Study Completion 2018-07-23 (Actual)

PRIMARY OUTCOMES:
Trial feasibility | 90 days
  Recruitment feasibility (recruitment rate)

SECONDARY OUTCOMES:
Vascular Event Rate [Safety and Tolerability] | Day 1, Day 4±1, day 90±7
  Number of participants with a vascular event (including limb ischaemia, recurrent stroke, myocardial infarction, venous thrombo-embolism)
Treatment Related Serious Adverse Event Rates [Safety and Tolerability] | Day 1, Day 4±1, day 90±7
  Number of participants with a serious adverse event related to treatment
Biomarkers | Immediately before RIC/sham at baseline; immediately after RIC/sham on Day 1; day 4±1
  Plasma S100-beta protein
Biomarkers | Immediately before RIC/sham at baseline; immediately after RIC/sham on Day 1; day 4±1
  Plasma heat-shock proteins
Biomarkers | Immediately before RIC/sham at baseline; immediately after RIC/sham on Day 1; day 4±1
  Plasma cytokines
Impairment | Day 4±1, day 90±7
  National Institutes of Health Stroke Scale
Dependency | Day 90±7
  Modified Rankin scale
Disability | Day 90±7
  Barthel Index
Mood | Day 90±7
  Zung depression scale
Telephone cognition | Day 90±7
  Modified Telephone Interview for Cognitive Status (TICS-M)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Derby Teaching Hospitals Foundation Trust, Derby, Derbyshire
  - Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] England TJ, Hedstrom A, O'Sullivan SE, Woodhouse L, Jackson B, Sprigg N, Bath PM. Remote Ischemic Conditioning After Stroke Trial 2: A Phase IIb Randomized Controlled Trial in Hyperacute Stroke. J Am Heart Assoc. 2019 Dec 3;8(23):e013572. doi: 10.1161/JAHA.119.013572. Epub 2019 Nov 21. PMID 31747864